CLINICAL TRIAL: NCT02645058
Title: Retrograde Intrarenal Surgery (RIRS) Versus Extracorporeal Shock Waves Lithotripsy (ESWL) for the Treatment of Renal Stones Measuring 6-20 mm: A Prospective Randomized Study
Brief Title: RIRS Versus ESWL for the Treatment of Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Ettore Dalmasso, Doctor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0016589
Record Dates: First submitted 2015-06-29; First posted 2016-01-01 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Renal Stones
Keywords: Ureterorenoscopy; extracorporeal shock waves lithotripsy
MeSH Terms: conditions — Nephrolithiasis | interventions — Lasers, Solid-State; Anesthesia, Spinal; Diagnostic Imaging; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIRS (retrograde intrarenal surgery) (Experimental): In the first arm (RIRS) the patients will be treated by a standard retrograde ureterorenoscopy and Holmium laser lithotripsy. Preoperative exams will be abdomen ultrasound and Xray (CT in case of stones > 15 mm), urine analysis and culture (according to all the more recent guidelines). Surgeries will be performed under general or spinal anesthesia, according to anesthesiologist evaluation. According with standard technique, ureteroscopy will be performed using both rigid and flexible ureteroscope. Lithotripsy will be performed by Holmium laser. Major stone fragments will be removed at the end of the procedure. Finally a double J ureteral stent will be push in specific cases depending on intraoperative findings (length of the procedure, macroscopic view of the ureter, residual stones etc.). RIRS will be an outpatients procedure with an hospital stay <23 hours. Some patients may require a longer hospital stay due to specific pre-operative diseases or intra/post-operative events.
  Interventions: Procedure: RIRS; Device: Rigid and flexible ureteroscope; Device: Holmium laser; Device: Basket for fragment removal; Procedure: General or spinal anesthesia; Device: X-ray
- ESWL (extracorporeal shockwaves lithotripsy) (Experimental): In the second arm (ESWL) the patients will be treated by a standard extracorporeal shock waves lithotripsy (ESWL). Preoperative exams will be the same as first arm. No general or spinal anaesthesia will be used, but just intravenous medications if required. Ultrasound and/or X-Ray will be used to locate the stone. Power and number of shock waves will consist in 20-24 KV and 3000-3500 sw respectively, according to individual tolerance. ESWL will be an outpatients procedure with an hospital stay <23 hours. Some patients may require a longer hospital stay due to specific pre-operative diseases or intra/post-operative events.
  Interventions: Procedure: ESWL; Device: Lithotripter; Drug: Intravenous pain medication; Device: X-ray; Device: Ultrasound

INTERVENTIONS:
Procedure: RIRS — Treatment by ureterorenoscopy (RIRS) and laser lithotripsy
  Arms: RIRS (retrograde intrarenal surgery)
Procedure: ESWL — Treatment by extracorporeal shock waves lithotripsy
  Arms: ESWL (extracorporeal shockwaves lithotripsy)
Device: Rigid and flexible ureteroscope
  Arms: RIRS (retrograde intrarenal surgery)
Device: Lithotripter
  Arms: ESWL (extracorporeal shockwaves lithotripsy)
Device: Holmium laser
  Arms: RIRS (retrograde intrarenal surgery)
Device: Basket for fragment removal
  Arms: RIRS (retrograde intrarenal surgery)
Procedure: General or spinal anesthesia
  Arms: RIRS (retrograde intrarenal surgery)
Drug: Intravenous pain medication — If required by the patient
  Arms: ESWL (extracorporeal shockwaves lithotripsy)
Device: X-ray — To focus the stone
Device: Ultrasound — To focus the stone
  Arms: ESWL (extracorporeal shockwaves lithotripsy)

SUMMARY:
To evaluate the effectiveness of RIRS (retrograde intrarenal surgery) and ESWL (extracorporeal shockwaves lithotripsy) in the treatment of renal stone ranging form 6 to 20 mm size.

DETAILED DESCRIPTION:
European urological guidelines consider RIRS and ESWL the treatments of choice for renal stones < 20 mm. RIRS is a endoscopic surgery which allows to rich the kidney from the ureter. A flexible ureteroscope is used for these kind of procedure. Through this device a laser fiber (Holmium laser) is used to treat the stones. After that, small fragments can be removed with a basket. In some cases, according to intraoperative findings, a ureteral stent can be push in the kidney to help the drainage of the kidney. ESWL is a procedure which allows to treat the stones by shock waves generated by a specific machine which work in direct contact with the skin of the patients (extracorporeal). Shockwaves pass all the tissues and finally reach the stones. Such energy allows to break the stones in small fragments, that wll be spontaneously passed by the patients. Specific parameters of these treatments are discussed in "Arms and Interventions". Many studies demonstrated high success rate of RIRS and this technique is becoming more and more adopt. One study demonstrated better outcomes of RIRS versus ESWL, but only for renal stones located in the inferior calices and smaller then 10 mm. There are not other studies comparing the two procedures and there are not proofs that RIRS ensures better outcomes for other renal stones (neither for size nor for location).

ELIGIBILITY:
Inclusion Criteria:

* renal stone measuring 6 to 20 mm
* signing informed consent
* WHO performance status 0-2

Exclusion Criteria:

* Other stone >5 mm
* concomitant ureteral stones
* BMI > 35
* severe coagulopathy
* impossibility to sign informed consent
* pregnancy
* age < 18 years old or > 85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Number of patients stone free SFR 4 | 1 month from treatment
  Patients with residual fragments < 5 mm after treatment

SECONDARY OUTCOMES:
Number of patients stone free SFR 0 | 1 month from treatment
  Patients with no residual fragments after treatment
Number of patients stone free SFR 4 | 6 months after the treatment
  Patients with residual fragments < 5 mm after treatment
Number of patients stone free SFR 0 | 6 months after the treatment
  Patients with no residual fragments after treatment
Number of patients stone free SFR 4 | 1 year after the treatment
  Patients with residual fragments < 5 mm after treatment
Number of patients stone free SFR 0 | 1 year after the treatment
  Patients with no residual fragments after treatment
rate of complications | within 1 month form treatment
  number of complications after treatment
rate of further treatment needed | within 1 year
  number of retreatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bosio, Medicine, Principal Investigator — Urology, University of Turin
Locations (1):
- Urology, University of Turin, Turin, Italy

REFERENCES:
- [Derived] Bosio A, Alessandria E, Dalmasso E, Agosti S, Vitiello F, Vercelli E, Bisconti A, Gontero P. Flexible Ureterorenoscopy Versus Shockwave Lithotripsy for Kidney Stones </=2 cm: A Randomized Controlled Trial. Eur Urol Focus. 2022 Nov;8(6):1816-1822. doi: 10.1016/j.euf.2022.04.004. Epub 2022 Apr 22. PMID 35466071